CLINICAL TRIAL: NCT02636920
Title: Study and Development of Application Models of "Therapeutic Education to the Patient" (TEP) in Asthmatic Children
Acronym: TEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stefania La Grutta, MD (Other)
Responsible Party: Sponsor-Investigator, Stefania La Grutta, MD, Stefania La Grutta, MD. Senior Researcher. Coordinator of Pediatric Allergy and Asthma Research Group. Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Organization: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 8/2014-
Record Dates: First submitted 2015-10-30; First posted 2015-12-22 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Asthma
Keywords: Asthma; Children
MeSH Terms: conditions — Asthma | interventions — tetraethylpyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEP-CASES (Other): 25 Case Patients will follow the Therapeutic Education to the Patient (TEP).
  In addition the following procedures will be performed:
  * Pediatric Asthma Quality of Life Questionnaire (PAQLQ);
  * Children Asthma Control Test (C-ACT);
  * Pediatric Caregiver Asthma Quality of Life Questionnaire (PCAQLQ);
  * Functional respiratory tests: forced expiratory volume in one second (FEV1), forced expiratory flow between 25% and 75% (FEF 25-75), forced vital capacity (FVC) and Peak expiratory flow (PEF)
  Interventions: Other: Therapeutic Education to the Patient (TEP)
- TEP-CONTROLS (No Intervention): 25 Control Patients will follow the usual care program:
  * The Pediatric Asthma Quality of Life Questionnaire (PAQLQ);
  * The Children Asthma Control Test (C-ACT);
  * the Pediatric Caregiver Asthma Quality of Life Questionnaire (PCAQLQ);
  * Functional respiratory tests: forced expiratory volume in one second (FEV1), forced expiratory flow between 25% and 75% (FEF 25-75), forced vital capacity (FVC) and Peak expiratory flow (PEF)

INTERVENTIONS:
Other: Therapeutic Education to the Patient (TEP) — * Educational Diagnosis, asking what patient has, what he knows, what he is doing, what he would like to do.
  * Therapeutic Contract, to define objectives to reach at the end of educational path, integrating new knowledges and replacing wrong cognitive-behavior models with new schemes.
  * Educational Therapeutic Intervention, with individual or group methodologies (Role Playing, Brain Storming) and a disease diary in which patients could describe symptoms, therapies, behaviors and benefits.
  * Assessing of the knowledges acquired by patients.
  Other Names: TEP
  Arms: TEP-CASES

SUMMARY:
It is an interventional prospective study. The study will assess the intervention of the "Therapeutic Education to the Patient (TEP)" on the quality of life in asthmatic children.

The patients will be enrolled from the 1st of May 2016 to the 31st of December 2016 in the outpatient clinic of Pediatric Allergology & Pulmonology (PAP) of Respiratory Disease Research Center (RDRC) within the Institute of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (RDRC-IBIM CNR), Italy.

DETAILED DESCRIPTION:
It is an interventional prospective study. The study will assess the intervention of the "Therapeutic Education to the Patient (TEP)" on the quality of life in asthmatic children.

The patients will be enrolled from the 1st of May 2016 to the 31st of December 2016 in the outpatient clinic of Pediatric Allergology & Pulmonology (PAP) of Respiratory Disease Research Center (RDRC) within the Institute of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (RDRC-IBIM CNR), Italy.

25 Case Patients will follow the Therapeutic Education to the Patient (TEP) and 25 Control Patients will follow the usual care program.

The following procedures will be performed:

* Pediatric Asthma Quality of Life Questionnaire (PAQLQ);
* Children Asthma Control Test (C-ACT);
* Pediatric Caregiver Asthma Quality of Life Questionnaire (PCAQLQ);
* Familiar Empowerment Scale (FES);
* Functional respiratory tests: forced expiratory volume in one second (FEV1), forced expiratory flow between 25% and 75% (FEF 25-75), forced vital capacity (FVC) and Peak expiratory flow (PEF); in addition, FEV1 and PEF will be daily recorded through the SmartOne device (Medical International Research s.r.l.), a portable flow peak meter for smartphones;
* Evaluation of the presence of Cotinine and Nicotine from Hair and Urine analysis respectively;
* Evaluation of levels of exposure to polycyclic aromatic hydrocarbons (PAH) through urine analysis.

Data collection about asthma control, quality of life and spirometry will be managed through DragONE, a downloadable APP for smartphones.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma

Exclusion Criteria:

* Acute respiratory infection signs
* Immunologic and metabolic systemic disease
* Major malformation of upper respiratory tract
* Active smokers patients

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Impact of a Short Early Therapeutic Education Program on Quality of life of asthmatic children | 2 YEARS
  The main objective is to measure the impact of the program on the QOL of asthmatic primary-school aged children seen for the first time in consultation with a pediatric pulmonologist.
  QOL of the children, will be assessed by Pediatric Asthma Quality of Life Questionnaire, PAQLQ.

SECONDARY OUTCOMES:
Impact of a Short Early Therapeutic Education Program on QOL of Parents of asthmatic children | 2 YEARS
  The secondary objective is to assess the effects of the program on the QOL of parents.
  QOL of the accompanying parent will be assessed by the Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ)
Impact of a Short Early Therapeutic Education Program on Asthma Management of asthmatic children | 2 YEARS
  The secondary objective is to assess the effects of the program on asthma management.
  Asthma management will be assessed by Childhood Asthma Control Test (C-ACT)
Impact of a Short Early Therapeutic Education Program on Functional respiratory test of asthmatic children | 2 YEARS
  The secondary objective is to assess the effects of the program on parameters of functional respiratory tests.(FRT).
  FRT will be assessed by forced expiratory volume in one second (FEV1), forced expiratory flow between 25% and 75% (FEF 25-75), the forced vital capacity (FVC) and Peak expiratory flow (PEF).
Presence of Cotinine and Nicotine from Hair and Urine analysis respectively | 2 YEARS
Levels of exposure to polycyclic aromatic hydrocarbons (PAH) through urine analysis | 2 YEARS

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Biomedicine and Molecular Immunology (IBIM), National Research Council, Palermo, Sicily, Italy